CLINICAL TRIAL: NCT01571336
Title: Non-interventional Observational Study on Photodynamic Therapy of Actinic Keratoses With Alacare®
Brief Title: Photodynamic Therapy of Actinic Keratoses With Alacare®
Status: Completed | Type: Observational
Sponsor: photonamic GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS 01
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to collect data on the frequency of SCCs in the Alacare®-treated area during an interval of two years after Alacare®-PDT.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients with 3 to 6 mild AK lesions on the hairless areas of the head and face which were treated with Alacare®-PDT according to the SPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2012-04; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of SCCs in areas treated with Alacare®-PDT | Two years after Alacare®-PDT

CONTACTS AND LOCATIONS:
Overall Officials: Peter Radny, MD, Study Chair — Dermatological group practice, Charlottenstraße 12, D-88045 Friedrichshafen, Germany
Locations (8):
- Germany (8):
  - Medizinisches Zentrum Bonn Friedensplatz, Bonn
  - Hautarztpraxis Prof. Kurzen, Freising
  - Hautärztliche Gemeinschaftspraxis Dr. med. Peter Dworzak Dr. med. Peter Radny, Friedrichshafen
  - Gemeinschaftspraxis Dres.Ina Röhrig-Petering und Holger Petering, Hildesheim
  - Dermatologische Gemeinschaftspraxis Prof. Dr. J. Gille & Dr. K. Spieth-Gille, Königstein im Taunus
  - ZENTderma, Mönchengladbach
  - Facharzt für Haut- und Geschlechtskrankheiten, Radolfzell
  - Praxis Prof. Dr. Thomas Dirschka, Wuppertal